CLINICAL TRIAL: NCT05093985
Title: Investigating the Effect of Neuromuscular Electrical Stimulation and Blood Flow Restriction Training on Physiological Deconditioning During Unloading and Retraining
Brief Title: Blood Flow Restricted Electrical Stimulation During Immobilisation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SMU-BFRImmob
Record Dates: First submitted 2021-09-20; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Atrophy, Muscular; Atrophy, Disuse
Keywords: immobilisation; blood flow restriction; neuromuscular electrical stimulation
MeSH Terms: conditions — Muscular Atrophy; Muscular Disorders, Atrophic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neuromuscular electrical stimulation with blood flow restriction (Experimental): This is the intervention condition
  Interventions: Other: Neuromuscular electrical stimulation with blood flow restriction
- No intervention (No Intervention): This is the control condition

INTERVENTIONS:
Other: Neuromuscular electrical stimulation with blood flow restriction — Neuromuscular electrical stimulation with blood flow restriction
  Arms: Neuromuscular electrical stimulation with blood flow restriction

SUMMARY:
Following injury or surgery to a limb, it is often immobilised to allow tissue healing. Short periods of disuse cause loss of muscle size and strength and impaired mechanical properties of tendons, which leads to reduced function. Strategies to combat these deconditioning adaptations include neuromuscular electrical stimulation (NMES), however at present its effectiveness is limited. Recent research suggests that the effects of NMES can be augmented with blood flow restriction (BFR). At present, the effect of combining these two techniques on muscle function during limb immobilisation is unknown. Furthermore, the impact of BFR training during retraining following immobilisation is unknown.

DETAILED DESCRIPTION:
Following injury or surgery to a limb, it is often immobilised to allow tissue healing. Short periods of disuse cause loss of muscle size and strength and impaired mechanical properties of tendons, which leads to reduced function. Strategies to combat these deconditioning adaptations include neuromuscular electrical stimulation (NMES), however at present its effectiveness is limited. Recent research suggests that the effects of NMES can be augmented with blood flow restriction (BFR). At present, the effect of combining these two techniques on muscle function during limb immobilisation is unknown. Furthermore, the impact of BFR training during retraining following immobilisation is unknown.

This study will examine the effectiveness and feasibility of a neuromuscular electrical stimulation and blood flow restriction protocol during a 7 day period of immobilisation. Multiple measures across several physiological systems will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 18-55
* Non-smoker
* No previous history of cardiovascular, respiratory or neurological problems
* Not taking anticoagulant medication
* Injury-free in the 3 months prior to scheduled participation in the study.

Exclusion Criteria:

* Hypertension (<140/80)
* Metal work in-situ
* Blood diseases or clotting issues
* Injury or previous injury (<3 months prior to scheduled participation in the study)
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in maximal isometric strength via Biodex Dynamometer | Through study completion, an average of 1 year
  Strength measure
Change in maximal isokinetic strength via Biodex Dynamometer | Through study completion, an average of 1 year
  Strength measure

SECONDARY OUTCOMES:
Change in muscle endurance via Biodex Dynamometer | Through study completion, an average of 1 year
  Endurance measure
Change in muscle morphology via 2D and 3D ultrasonography | Through study completion, an average of 1 year
  Morphology measure
Change in muscle VO2 via near-infrared spectroscopy | Through study completion, an average of 1 year
  VO2 measure
Change in blood markers via venous blood samples | Through study completion, an average of 1 year
  Blood markers
Change in pressure pain thresholds via handheld allometry | Through study completion, an average of 1 year
  Pain measure
Change in corticomotor excitability and inhibition, via transcranial magnetic stimulation | Through study completion, an average of 1 year
  Corticospinal function

IPD SHARING:
Plan to Share IPD: No